CLINICAL TRIAL: NCT03399799
Title: A Phase 1, First-in-Human, Open-Label, Dose Escalation Study of Talquetamab, a Humanized GPRC5D x CD3 Bispecific Antibody, in Subjects With Relapsed or Refractory Multiple Myeloma
Brief Title: Dose Escalation Study of Talquetamab in Participants With Relapsed or Refractory Multiple Myeloma
Acronym: MonumenTAL-1
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CR108404; 64407564MMY1001 (Other: Janssen Research & Development, LLC); 2017-002400-26 (EudraCT Number); 2023-504581-29-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2017-12-22; First posted 2018-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Hematological Malignancies
MeSH Terms: conditions — Hematologic Neoplasms | interventions — talquetamab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: Dose Escalation (Talquetamab) - Intravenous (IV) (Experimental): Participants will receive IV infusion of Talquetamab at minimum anticipated biologic effect level (MABEL)-based starting dose until the completion of the end of treatment visit. Subsequent dose levels will be selected based on the review of all available data including, but not limited to, pharmacokinetic, pharmacodynamic, safety, and preliminary antitumor activity data. Participants receiving IV dosing can transition to SC dosing through-out the study upon sponsor consultation. All participants (ongoing and those who are in follow-up) will transition to open-label extension (OLE) phase and will continue to receive the study treatment. Upon approval of amendment 19 and notification from the sponsor, participants will transition to the long-term extension (LTE) and will continue to receive study treatment.
  Interventions: Drug: Talquetamab
- Part 1: Dose Escalation (Talquetamab) - Subcutaneous (SC) (Experimental): Participants will receive Talquetamab SC. The dose levels will be selected to identify safe and tolerable putative RP2D(s). All participants (ongoing and those who are in follow-up) will transition to OLE phase and will continue to receive the study treatment. Upon approval of amendment 19 and notification from the sponsor, participants will transition to the LTE and will continue to receive study treatment.
  Interventions: Drug: Talquetamab
- Part 2: Dose Expansion (Talquetamab) (Experimental): Participants will receive IV infusion or SC injection of Talquetamab at each putative recommended Phase 2 dose(s) (RP2D[s]) as determined in Part 1. Participants receiving IV dosing can transition to SC dosing through-out the study upon sponsor consultation. All participants (ongoing and those who are in follow-up) will transition to OLE phase and will continue to receive the study treatment. Upon approval of amendment 19 and notification from the sponsor, participants will transition to the LTE and will continue to receive study treatment.
  Interventions: Drug: Talquetamab

INTERVENTIONS:
Drug: Talquetamab — Participants will receive IV infusion or SC injection of Talquetamab.

SUMMARY:
The purpose of this study is to characterize the safety of Talquetamab and to determine the recommended Phase 2 dose(s) (RP2Ds) and dosing schedule assessed to be safe for Talquetamab (Part 1 [Dose Escalation]) and to further characterize the safety of Talquetamab at the recommended Phase 2 dose(s) (RP2Ds) (Part 2 [Dose Expansion]).

ELIGIBILITY:
Inclusion Criteria:

* Documented initial diagnosis of multiple myeloma according to International Myeloma Working Group (IMWG) diagnostic criteria
* Part 1: Participants with measurable multiple myeloma who have progressed on, or could not tolerate, all available established therapies. Part 2: Participants with multiple myeloma measurable by central laboratory assessment who have progressed on, or could not tolerate, all available established therapies; Serum monoclonal paraprotein (M-protein) level greater than or equal to (>=) 1.0 gram per deciliter (g/dL) or urine M-protein level >=200 milligram per 24 hours (mg/24 h) or light chain multiple myeloma without measurable disease in the serum or the urine: serum immunoglobulin free light chain (FLC) >= 10 mg/dL and abnormal serum immunoglobulin kappa lambda FLC ratio; If central laboratory assessments are not available, relevant local laboratory measurements must exceed the minimum required level by at least 25%
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1
* Women of childbearing potential must have a negative pregnancy test at screening and prior to the first dose of study drug using a highly sensitive pregnancy test either serum (Beta human chorionic gonadotropin [beta-hCG]) or urine
* Sign an informed consent form (ICF) indicating that he or she understands the purpose of and procedures required for the study, and is willing to and able participate in the study. Consent is to be obtained prior to the initiation of any study-related tests or procedures that are not part of standard-of-care for the participant's disease

Exclusion Criteria:

* Participants who received or plan to receive any live, attenuated vaccine within 4 weeks prior to the first dose, during treatment, or within 4 weeks of the last dose of Talquetamab. Non-live or non-replicating vaccines approved or authorized for emergency use (example, coronavirus disease [COVID]-19) by local health authorities are allowed
* Toxicities from previous anticancer therapies should have resolved to baseline levels or to Grade 1 or less except for alopecia or peripheral neuropathy
* Received a cumulative dose of corticosteroids equivalent to greater than or equal to ( >=) 140 milligram (mg) of prednisone within the 14-day period before the first dose of study drug (does not include pretreatment medication)
* An allogenic stem cell transplant within 6 months before first dose of study drug. Participants who received an allogeneic transplant must be off all immunosuppressive medications for 6 weeks without signs of graft-versus-host disease (GVHD); and/or an autologous stem cell transplant less than or equal to (<=) 12 weeks before first dose of study drug
* Documented history of central nervous system (CNS) involvement or exhibits clinical signs of meningeal involvement of multiple myeloma. If either is suspected, whole body magnetic resonance imaging (MRI) and lumbar cytology are required

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2017-12-16 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2029-03-30 (Estimated)

PRIMARY OUTCOMES:
Part 1: Dose-limiting Toxicity (DLT) | Up to Day 28
  The Dose Limiting Toxicities (DLTs) are based on drug related adverse events and defined as any of the following events: hematological / non-hematological toxicity of Grade 3 or higher.
Part 1 and Part 2: Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | From signing of Informed Consent Form (ICF) up to follow up (until 100 days after the last dose of study drug or until the start of subsequent anticancer therapy, if earlier [approximately 2.10 years])
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.

SECONDARY OUTCOMES:
Part 1: Talquetamab Serum Concentrations | Up to 4 weeks
  Serum concentrations will be calculated for Talquetamab.
Part 1 and Part 2: Biomarker Assessment | Up to Cycle 7 Day 1 (each cycle of 21-days)
  Serum cytokine concentrations will be measured pre- and post-infusion of Talquetamab for biomarker assessment.
Part 1: Number of Participants with Talquetamab Antibodies | Up to 4 weeks
  Antibodies to Talquetamab will be assessed to evaluate potential immunogenicity.
Part 2: Overall Response Rate (ORR) | Approximately 2.10 years
  ORR is defined as the proportion of participants who have a partial response (PR) or better according to the international myeloma working group (IMWG) criteria.
Part 2: Clinical Benefit Rate (CBR) | Approximately 2.10 years
  CBR is defined as the proportion of participants who have a minimal response (MR) or better according to the IMWG criteria.
Part 2: Duration of Response (DOR) | From the date of initial documentation of a response to the date of first documented evidence of progressive disease (PD) (approximately 2.10 years)
  DOR is defined as time from date of initial documentation of a response (PR or better) to date of first documented evidence of PD, per IMWG criteria.
Part 2: Time to Response (TTR) | From the date of first dose of study drug to the date of initial documentation of a response (approximately 2.10 years)
  TTR is defined as the time between date of first dose of study drug and the first efficacy evaluation that the participant has met all criteria for PR or better.
Part 2: Progression-Free Survival (PFS) | Every 16 weeks until end of study, participant dies, withdrawn consent, or lost to follow up (up to 18 months)
  PFS is defined as time from date of first dose of study drug to date of first documented PD, per IMWG criteria, or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (13):
- United States (5):
  - University of Alabama Birmingham, Birmingham, Alabama
  - City of Hope, Duarte, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Mount Sinai Medical Center, New York, New York
  - Tennessee Oncology, Nashville, Tennessee
- Centre Hospitalier Universitaire de Liege Domaine Universitaire du Sart Tilman, Liège, Belgium
- Netherlands (2):
  - VU Medisch Centrum, Amsterdam
  - UMCU, Utrecht
- Spain (5):
  - Hosp. Univ. Germans Trias I Pujol, Badalona
  - Hosp Univ Fund Jimenez Diaz, Madrid
  - Clinica Univ. de Navarra, Pamplona
  - Hosp. Quiron Madrid Pozuelo, Pozuelo de Alarcón
  - Hosp Clinico Univ de Salamanca, Salamanca

REFERENCES:
- [Derived] Einsele H, Moreau P, Bahlis N, Bhutani M, Vincent L, Karlin L, Perrot A, Goldschmidt H, van de Donk NWCJ, Ocio EM, Martinez Lopez J, Rodriguez-Otero P, Dytfeld D, Jakubowiak A, Schinke C, Besemer B, Anguille S, Manier S, Rasche L, Teipel R, Scheid C, Pawlyn C, Cavo M, Diels J, Ghilotti F, Lau BW, Renaud T, Orel O, Ong F, Ramos DF, Ammann E, Parekh T, Albrecht C, Weisel K, Mateos MV. Comparative Efficacy of Talquetamab vs. Real-World Physician's Choice of Treatment in Triple-Class-Exposed Relapsed/Refractory Multiple Myeloma: Updated Analyses of MonumenTAL-1 vs. LocoMMotion/MoMMent. Adv Ther. 2025 Nov 28. doi: 10.1007/s12325-025-03409-y. Online ahead of print. PMID 41313549
- [Derived] Schinke C, Rodriguez-Otero P, van de Donk NWCJ, Lipe B, Lavi N, Rasche L, Parekh S, Van Oekelen O, Vishwamitra D, Skerget S, Cortes-Selva D, Verona R, Hilder B, Masterson T, Campagna M, Khedkar S, Renaud T, Tolbert J, Kane C, Gray KS, Saber I, Heuck C, Chari A. Infections and parameters of humoral immunity with talquetamab in relapsed/refractory multiple myeloma in MonumenTAL-1. Blood Adv. 2025 Nov 25;9(22):5752-5762. doi: 10.1182/bloodadvances.2025016613. PMID 40864183
- [Derived] Schinke C, Touzeau C, Oriol A, Mateos MV, Stevens D, Rasche L, Qin X, Kato K, Bathija S, Katz EG, Gries KS, Campagna M, Masterson T, Hilder BW, Tolbert J, Renaud T, Heuck C, Tomlinson C, Moreau P, San-Miguel J, Rodriguez-Otero P, Chari A. Talquetamab improves patient-reported symptoms and health-related quality of life in relapsed or refractory multiple myeloma: Results from the phase 1/2 MonumenTAL-1 study. Cancer. 2025 Jul 15;131(14):e35927. doi: 10.1002/cncr.35927. PMID 40631904
- [Derived] Chari A, Touzeau C, Schinke C, Minnema MC, Berdeja JG, Oriol A, van de Donk NWCJ, Rodriguez-Otero P, Morillo D, Martinez-Chamorro C, Mateos MV, Costa LJ, Caers J, Rasche L, Krishnan A, Ye JC, Karlin L, Lipe B, Vishwamitra D, Skerget S, Verona R, Ma X, Qin X, Ludlage H, Campagna M, Masterson T, Hilder B, Tolbert J, Renaud T, Goldberg JD, Kane C, Heuck C, San-Miguel J, Moreau P. Safety and activity of talquetamab in patients with relapsed or refractory multiple myeloma (MonumenTAL-1): a multicentre, open-label, phase 1-2 study. Lancet Haematol. 2025 Apr;12(4):e269-e281. doi: 10.1016/S2352-3026(24)00385-5. Epub 2025 Mar 13. PMID 40090350
- [Derived] Catamero D, Ray C, Purcell K, Leahey S, Esler E, Rogers S, Hefner K, O'Rourke L, Gray K, Tolbert J, Renaud T, Patel S, Hannemann L, Shenoy S. Nursing Considerations for the Clinical Management of Adverse Events Associated with Talquetamab in Patients with Relapsed or Refractory Multiple Myeloma. Semin Oncol Nurs. 2024 Oct;40(5):151712. doi: 10.1016/j.soncn.2024.151712. Epub 2024 Aug 17. PMID 39155155
- [Derived] Chari A, Minnema MC, Berdeja JG, Oriol A, van de Donk NWCJ, Rodriguez-Otero P, Askari E, Mateos MV, Costa LJ, Caers J, Verona R, Girgis S, Yang S, Goldsmith RB, Yao X, Pillarisetti K, Hilder BW, Russell J, Goldberg JD, Krishnan A. Talquetamab, a T-Cell-Redirecting GPRC5D Bispecific Antibody for Multiple Myeloma. N Engl J Med. 2022 Dec 15;387(24):2232-2244. doi: 10.1056/NEJMoa2204591. Epub 2022 Dec 10. PMID 36507686
- [Derived] Pillarisetti K, Edavettal S, Mendonca M, Li Y, Tornetta M, Babich A, Majewski N, Husovsky M, Reeves D, Walsh E, Chin D, Luistro L, Joseph J, Chu G, Packman K, Shetty S, Elsayed Y, Attar R, Gaudet F. A T-cell-redirecting bispecific G-protein-coupled receptor class 5 member D x CD3 antibody to treat multiple myeloma. Blood. 2020 Apr 9;135(15):1232-1243. doi: 10.1182/blood.2019003342. PMID 32040549
- See also: A Study of Talquetamab in Participants With Relapsed or Refractory Multiple Myeloma — https://clinicaltrials.gov/ct2/show/NCT04634552